CLINICAL TRIAL: NCT06505460
Title: Exploring the Possible Beneficial Impact of Non-invasive and Invasive Neuromodulation on Freezing of Gait in Parkinson's Disease During Different Ambulatory Complexities: An Electrophysiological and fMRI Study
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: China Medical University Hospital (Other)
Collaborators: Ministry of Science and Technology, Taiwan (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CMUH112-REC2-213
Record Dates: First submitted 2024-07-11; First posted 2024-07-17 (Actual); Last update posted 2024-08-21 (Actual); Status verified 2024-08

CONDITIONS: Transcranial Direct Current Stimulation
Keywords: Parkinson's disease; freezing of gait; MRI; tDCS; focused ultrasound; DBS
MeSH Terms: conditions — Parkinson Disease | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- real tDCS (Experimental): In transcranial direct current stimulation, the constant current of 2.0 mA was applied to each site for up to 20 minutes.
  Interventions: Device: Transcranial direct current stimulation
- sham tDCS (Sham Comparator): In transcranial direct current stimulation, the sham stimulation will be 30s stimulation with ramp up and ramp off for 10s at 2.0 mA.
  Interventions: Device: Transcranial direct current stimulation

INTERVENTIONS:
Device: Transcranial direct current stimulation — A consecutive 5-days course of tDCS will be delivered. In treatment group, true stimulation will be administrated and sham stimulation will be delivered in control group.

SUMMARY:
Freezing of gait (FOG) stands out as a devastating symptom of Parkinson's disease (PD), where patients may become momentarily glued to the ground, rendering them incapable of walking efficiently. The pathogenesis of FOG remains uncertain but is likely attributed to functional perturbations in superficial cortical and deep locomotion regions. FOG tends to manifest more prominently during complex walking, such as turning, than during simple straight forward walking, and the reasons for this phenomenon remain unclear. Unfortunately, effective methods for overcoming this ambulatory issue has yet to be identified, and quantifying paroxysmal gait spells proves challenging with clinical rating alone; thus, a scientific tool is warranted. In this 3-year proposal, the investigators plan to address these challenges comprehensively.

DETAILED DESCRIPTION:
First, the investigators aim to develop an artificial intelligence algorithm for the identification and quantification of FOG episodes using Red-Green-Blue (RGB) and walkway pressure data. PD patients experiencing FOG will undergo a standardized walking protocol on the PKMAS System, acquiring simultaneous data from two angles of video recording and foot pressure. Labeled videos of FOG incidents will be inputted into an algorithm, Adaptive Fusion Algorithm for Spam Detection (AFSD), utilizing raw RGB data, optical flow data (DualTVL), and their combination for temporal segmentation.

Second, the investigators intend to pinpoint sources of FOG in PD patients through electrophysiological methods during unconstrained walking, employing a high-density 64-channel electroencephalographic ambulatory recording and motor imagery fMRI to delve into the pathophysiology of FOG under different ambulatory conditions. Effective connectivity among higher neural regions, including the basal ganglia, cerebellum, and cortical regions, will be explored. The resulting connectivity map will be overlaid with electric recording data to examine neurovascular coupling or uncoupling.

Third, the investigators plan to conduct non-invasive interventions (transcranial direct current stimulation: tDCS, magnetic resonance-guided focused ultrasound: MRgFUS) and Deep Brain Stimulation (DBS) to assess their impact on gait and FOG in PD patients. Motor imagery fMRI and electrophysiological investigations will be performed before and after treatment using the mentioned methods. Our multi-modal approach aims to unravel the complexities of FOG in PD patients, providing valuable insights and potentially benefiting those enduring the challenges posed by this debilitating symptom.

ELIGIBILITY:
Inclusion Criteria:

1. Patients meet the diagnosis of PD based on the established consensus criteria
2. Age above 20 years old and below 90 years
3. For MRgFUS patients: a. At least one of the 3 cardinal symptoms (akinesia, tremor, rigidity) reaches an intensity of at least 2/4. b. Parkinsonian symptoms cannot be satisfactorily controlled by optimal pharmacological treatment including L-dopa and other antiparkinsonian drugs. c. stable medication for PD ≥ 30 days.
4. DBS patients must meet Taiwan Health Insurance criteria: PD duration exceeding 5 years, positive response to levodopa (≥33% UPDRS motor score improvement), and presence of motor complications (e.g., wearing off, on-off, levodopa-related dyskinesia, or medically intractable tremor).

Exclusion Criteria:

1. Congestive heart failure (Functional III or above) or advanced cancer with distant metastasis.
2. PD at Hoehn and Yahr Stage 5.
3. DBS exclusion criteria: overt dementia or major depression.

Ages: 20 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-04-30 (Actual); Primary Completion 2025-07-31 (Estimated); Study Completion 2027-07-31 (Estimated)

PRIMARY OUTCOMES:
Electroencephalogram recording before and after the tDCS session | baseline / 2 days, 2 and 4 weeks after the end of the tDCS session
  Gait recording by 64 channels EEG device. Four different frequency bands ( theta, alpha, beta, and gamma) will be investigated. Variables in gait analysis: 1.Gait initiation, 2.Level walking, 3.Gait termination.
Electromyography recording before and after the tDCS session | baseline / 2 days, 2 and 4 weeks after the end of the tDCS session
  The 4 pairs of leg EMG recording during 50 meters walking. The EMG signals will be filtered with a band pass ranging from 0.05 to 70 Hz. Variables in gait analysis: 1.Gait initiation, 2.Level walking, 3.Gait termination.
Functional magnetic resonance images examination before and after the tDCS session | baseline / 2 days after the end of the tDCS session
  fMRI scan will be performed on a 3.0T MR imager to detect the brain BOLD signal change in FOG. When fMRI was conducted, four different video tapes will be presented to the subjects#1.normal walking, 2.normal turning, 3.FOG during forward straight walking and 4.FOG during turning.
Change in Unified Parkinson's Disease Rating Scale (UPDRS) Part III before and after the tDCS session UPDRS contains four parts, the third part of which is reported in this outcome. | baseline / 2 days, 2 and 4 weeks after the end of the tDCS session
  UPDRS contains four parts, the third part of which is reported in this outcome. Part III is clinician-scored monitored motor evaluation (14 questions, ranges from 0=normal to 4= Severe). The scoring of Part III varies between 0-56. The higher score indicates the worse motor function. Negative change from baseline values indicate improvement.

SECONDARY OUTCOMES:
Change in New freezing of gait questionnaire (NFOG-Q) before and after the tDCS session | baseline / 2 days, 2 and 4 weeks after the end of the tDCS session
  NFOG-Q contains three parts: in the first part, a video clip will be shown to the participants with PD and help to classify whether an individual is a freezer or non-freezer. The second and third part of the questionnaire is designed for freezers only. Par II (items 2-6, scores range between 0-19) assesses the severity of FOG according to the frequency and duration of the freezing episodes. Part III (items 7-9, scores range between 0-9) evaluates the impact of freezing on daily activities. The higher score indicates the worse freezing of gait. Negative change from baseline values indicate improvement.
Change in Gait and Falls Questionnaire (GFQ) before and after the tDCS session | baseline / 2 days, 2 and 4 weeks after the end of the tDCS session
  Gait and Falls Questionnaire assesses freezing of gait severity in patients with Parkinson's Disease (16 questions, ranges from 0=normal to 4= Severe). The scoring varies between 0-64. The higher score indicates the worse motor function. Negative change from baseline values indicate improvement.

OTHER OUTCOMES:
Change in Tinetti's Mobility Index total score before and after the tDCS session | baseline / 4 weeks after the end of the tDCS session
  The Tinetti's Mobility Index contains two parts, Part I is Balance tests (9 questions, scores range between 0-16) and Part II is Gait tests (7 questions, scores range between 0-12). The scoring of this scale varies between 0 and 28 (< 19 high fall risk, 19-24 medium fall risk, 25-28 low fall risk). Positive change from baseline values indicate improvement.
Change in Berg Balance Scale before and after the tDCS session | baseline / 4 weeks after the end of the tDCS session
  Berg Balance Scale is clinician-scored monitored motor evaluation (14 questions, ranges from 0=normal to 4= Severe). The scoring varies between 0-56. The higher score indicates the worse motor function. Negative change from baseline values indicate improvement.
Change inParkinson's Disease Questionnaire 39 (PDQ-39) before and after the tDCS session | baseline / 4 weeks after the end of the tDCS session
  PDQ-39 is composed of 39 questions, divided into 8 parts: mobility, activities of daily living (ADLs), emotional wellbeing, stigma, social support, cognition, communication and physical discomfort. It assesses how often people affected by Parkinson's experience difficulties across 8 dimensions of daily living. All questions range from 0 to 4 (0=never, 4=always). The scoring of this scale varies between 0-156. Negative change from baseline values indicate better quality of life rating.
Non-Motor Symptoms Questionnaire (NMSQ) | baseline / 4 weeks after the end of the tDCS session
  Non-Motor Symptoms Scale for Parkinson's Disease is composed of 30 questions, divided into 9 parts: Cardiovascular including falls, Sleep/fatigue, Mood/cognition, Perceptual problems/hallucinations, Attention/memory, Gastrointestinal tract, Urinary, Sexual function and Miscellaneous. The scoring method is frequency x severity (higher scores = more disability, lower scores = less disability). Negative change from baseline values indicate improvement.

CONTACTS AND LOCATIONS:
Locations (1):
- China Medical University Hospital/Neuro Depart, Taichung, Taiwan